CLINICAL TRIAL: NCT03025945
Title: Pseudophakic Cystoid Macular Edema Prevention and Risk Factors; Prospective Study With Adjunctive Once Daily Topical Nepafenac 0.3% Versus Placebo
Brief Title: Prospective Study With Adjunctive Once Daily Topical Nepafenac 0.3% Versus Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intuor Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CME and nepafenac 0.3%
Record Dates: First submitted 2017-01-14; First posted 2017-01-20 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Cystoid Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- nepafenac 0.3% (Experimental): nepafenac 0.3% ophthalmic solution dosed once daily
  Interventions: Drug: Nepafenac 0.3%
- Saline Solution (Placebo Comparator): sterile saline drops with a pH approximately of 7.0 and osmolality of 290 mOsm/kg, dosed at once daily
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Nepafenac 0.3%
  Arms: nepafenac 0.3%
Drug: Saline Solution
  Arms: Saline Solution

SUMMARY:
Prospective, randomized, double-masked, placebo-controlled clinical study to define the effective use of a topical non-steroidal anti-inflammatory drug added to topical steroid use after uncomplicated phacoemulsification for the prevention of pseudophakic cystoid macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, 18 and older subjects with visually significant cataracts and were to undergo phacoemulsification with implantation of an intracapsular positioned intraocular lens.

Exclusion Criteria:

* previous uveitis (<1 year) previous anterior segment intraocular surgery hypersensitivity or allergy to NSAIDs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2013-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean McCafferty, MD, Principal Investigator — Arizona Eye Consultants

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCafferty S, Harris A, Kew C, Kassm T, Lane L, Levine J, Raven M. Pseudophakic cystoid macular edema prevention and risk factors; prospective study with adjunctive once daily topical nepafenac 0.3% versus placebo. BMC Ophthalmol. 2017 Feb 20;17(1):16. doi: 10.1186/s12886-017-0405-7. PMID 28219426

RESULTS

PARTICIPANT FLOW:
Groups:
- Nepafenac 0.3%: nepafenac 0.3% ophthalmic solution dosed once daily
  Nepafenac 0.3%
- Saline Solution: sterile saline drops with a pH approximately of 7.0 and osmolality of 290 mOsm/kg, dosed at once daily
  Saline Solution
Period: Overall Study
Arm/Group | Nepafenac 0.3% | Saline Solution
Started | 331 | 331
Completed | 331 | 331
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Six hundred and sixty two (662) patients, one thousand eyes (1000), completed the study. 1:1 ratio of control: treatment. Subjects were chosen from patients who had visually significant cataracts and were to undergo phacoemulsification with implantation of an intracapsular positioned intraocular lens.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Nepafenac 0.3% | Saline Solution | Total
Number analyzed (Participants) | 331 | 331 | 662
Number analyzed (Eyes) | 500 | 500 | 1000
Age, Continuous [Mean (Full Range); unit: years] | 68.8 [31 to 94] | 67.9 [39 to 96] | 68.3 [31 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 182 | 364
  Male | 149 | 149 | 298
Macular volume [Mean (Standard Deviation); unit: mm] | 8.7 (0.15) | 8.75 (0.15) | 8.72 (0.15)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Clinical Findings of Cystoid Macular Edema
Description: post-operative macular volume (mm)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Nepafenac 0.3% | Saline Solution
Number analyzed (Participants) | 331 | 331
Number analyzed (Eyes) | 500 | 500
mm | 8.85 (0.13) | 8.95 (0.18)

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Nepafenac 0.3% | Saline Solution
Serious Adverse Events (participants affected / at risk) | 0/331 | 0/331
Other Adverse Events (participants affected / at risk) | 1/331 | 0/331
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nepafenac 0.3% (N=331) | Saline Solution (N=331)
drop intolerance (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No